CLINICAL TRIAL: NCT04017299
Title: Choose an Electronic Distraction, Faisability and Discomfort Improvement Evaluation by and for ICU Patients : a Cross Over Randomized Controlled Study.
Brief Title: Electronic Distraction for ICU Patients
Acronym: CHOISIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL18_0218
Record Dates: First submitted 2019-07-05; First posted 2019-07-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Adult ICU Patients
Keywords: ICU; Pain; Anxiety; Thirst; Dyspnea; Sleep; Discomfort; Distress; Virtual Reality; Music Therapy
MeSH Terms: conditions — Pain; Anxiety Disorders; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Virtual reality with computer graphics (Active Comparator): Use of Virtual reality with computer graphics
  Interventions: Other: CHOISIR
- Virtual reality with real movies (Active Comparator): Use of Virtual reality with real movies
  Interventions: Other: CHOISIR
- Music therapy (dedicated device and music scores) (Active Comparator): Use of music therapy (dedicated device and music scores)
  Interventions: Other: CHOISIR
- Usual device (TV radio) (Other): usual distraction : watching TV
  Interventions: Other: CHOISIR

INTERVENTIONS:
Other: CHOISIR — Every patient will evaluate each device after 15 minutes of distraction once or twice a day according to the patient's wishes.

SUMMARY:
This is a feasibility study of electronic devices in order to reduce neuro-psychological disorders and suffering in intensive care unit (ICU) patients. A first step study is necessary to define which device is effective and safe to reduce symptom intensities, among music therapy, virtual reality with real pictures, virtual reality with artificial pictures, and common devices (radio or television). If some devices are effective to reduce patients' symptoms, a second step will be to implement and assess the impact of these tools in a multicenter trial.

DETAILED DESCRIPTION:
Quality of life following intensive care unit discharge is more and more anticipated during the ICU stay. Psychological trauma during ICU stay, related to medical management, can be very deleterious at short and long term, inducing psychological troubles as post-traumatic stress disorder and delaying the return to a normal social and professional life. For this reason, managing patients' distress is particularly important in the intensive care setting. There has been an increasing number of new technologies for the distraction of patients in different settings. a Today, a large amount of electronic distraction is available. TV and radio are available in each ICU, music therapy has already been studied and it is currently used in some ICUs. Virtual reality (VR) is used to improve attention and memory in stroke patients. Furthermore, VR seems to decrease stress post trauma disorders and phobia, as well as pain and anxiety during surgical procedures and physiotherapy. Our first step study will help us to determine which electronic distraction has the most effect on the top five discomfort symptoms frequently observed in ICU: pain, anxiety dyspnea, thirst and sleep privation.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted in intensive care unit,
* adult,
* French speaking,
* awake (RASS ≥ -1),
* not delirious (CAM-ICU negative),

Exclusion Criteria:

* patient refusal
* psychosis or preexisting cognitive dysfunction
* cerebral injury,
* hygiene/microbiological harm,
* pregnancy,
* decision of withdrawal of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Variation of intensity of the 5 discomfort symptoms (pain, anxiety, thirst, dyspnea, insomnia) assessed by a self-report 0-10 visually enlarged numeric rating scale | Just after the use of each device (up to 20 minutes)

SECONDARY OUTCOMES:
Variation of physiologic parametres (Heart Rate, Blood pressure, Respiratory rate and Analgesia nociception Index), evaluation of feasibility and feelings concerning the distraction devices. | ICU discharge (up to Day 28)
Variation of Respiratory rate during the use of each device | up to 20 minutes (after the device use )
  Respiratory rate : c/min
Variation of physiologic Blood pressure during the use of each device | up to 20 minutes (after the device use )
  Blood pressure : mmHg
Variation of Heart Rate during the use of each device | up to 20 minutes (after the device use )
  Heart Rate : b/min
evaluation of feasibility assessed by the Numeric Rating Scale from 0 to 10 | just after the use of each device (up to 20 minutes)
  Numeric Rating Scale from 0 to 10
Evaluation of the feelings concerning the distraction devices assessed by the Numeric Rating Scale from 0 to 10 | ICU discharge or up to Day 28
  Numeric Rating Scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Gérald CHANQUES, PhD, Principal Investigator — University of Montpellier Hospitals
Locations (1):
- University of Montpellier Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
identified data used in the published manuscript will be shared in accordance with the applicable informed consent under which the data was collected
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and IRB review. Dataset will be shared after careful examination by the study board of investigators.